CLINICAL TRIAL: NCT05050045
Title: Echocardiographic Screening of Healthy Neonates for Measuring Pulmonary Artery Pressure
Status: Completed | Type: Observational
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0106488
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Hypertension of Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present prospective study was to evaluate dynamic changes in both pulmonary artery pressure and ductus arteriosus during the first 72 hours after birth.

DETAILED DESCRIPTION:
Healthy newborn infants born in Alexandria University Children's Hospital were studied. Dynamic changes during the first 72 hours after birth were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 37-42 weeks.
* Birthweight: 2500-4000 g.

Exclusion Criteria:

* Neonates more than 6 hours of age at time of enrollment.
* Perinatal asphyxia or hypoxia (1 min Apgar scoring<7 points)
* Cardiac structural abnormalities detected by echocardiography except patent foramen ovale and patent ductus arteriosus
* Other clinically detected congenital malformations such as cleft lip and palate, omphalocele, meningocele, etc.
* Maternal history of gestational hypertension, gestational diabetes, hyperthyroidism, hypothyroidism, and autoimmune disease

Ages: 0 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy newborn infants born in Alexandria University Children's Hospital were studied. Dynamic changes in both pulmonary artery pressure and ductus arteriosus during the first 72 hours after birth were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery pressure (PAP) assessment - Tricuspid valve regurgitation peak velocity | up to 72 hours
  This is measured in apical 4 chamber view, with continuous wave Doppler using modified Bernoulli equation. Systolic pulmonary artery pressure is equivalent to right ventricular systolic pressure in absence of outflow obstruction.
  Systolic Pulmonary Artery Pressure (SPAP) = Right Ventricular Systolic Pressure = 4x TR2 + Right Atrial Pressure (RAP) (RAP= 3-5 mmHg)
Pulmonary artery pressure (PAP) assessment - Pulmonary regurgitation peak velocity | up to 72 hours
  This is measured in short axis parasternal view with continuous wave Doppler using this equation: Mean Pulmonary Artery Pressure MPAP= 4xPR2 + Right Ventricular Diastolic Pressure (RVdP=2-5 mmHg)
Pulmonary artery pressure (PAP) assessment - Transductal right-to-left flow peak velocity | up to 72 hours
  This is measured in high short axis ductal view with continuous wave Doppler
Pulmonary artery pressure (PAP) assessment - Interventricular septum configuration | up to 72 hours
  This is measured in short axis parasternal view above level of papillary muscles, left ventricle is normally O shaped, D or crescent shape indicated bowing of septum due to RV dysfunction.
Pulmonary artery pressure (PAP) assessment - Left ventricle systolic eccentricity index (LV-sEI) | up to 72 hours
  This is measured in short axis parasternal view by measuring LV dimensions the parallel versus the perpendicular dimension. The normal ratio is 1.
Right ventricular performance - Tricuspid annular plane systolic excursion(TAPSE) | up to 72 hours
  This is measured using Mmode in apical 4 chamber view over lateral annulus of tricuspid valve
Right ventricular performance - Myocardial Performance Index (MPI) | up to 72 hours
  This is measured by using pulsed wave doppler to measure isovolumetric ejection time + isovolumetric relaxation time/ right ventricular ejection time.
Right ventricular performance - E/A ratio | up to 72 hours
  This is measured in apical 4 chamber view by pulsed wave Doppler on mitral valve. The cut off value: 0.8- 2.
Left ventricular performance - Ejection fraction | up to 72 hours
  This is measured using M-Mode in long axis parasternal view with a normal range of 55-75%
Left ventricular performance - E/A ratio | up to 72 hours
  This is measured in apical 4 chamber view by pulsed wave Doppler on mitral valve. The cut off value: 0.8- 2
Shunts evaluation - Patent Ductus arteriosus | up to 72 hours
  Size will be evaluated in short axis parasternal view
Shunts evaluation - Patent Ductus arteriosus | up to 72 hours
  Direction will be evaluated in short axis parasternal view using color Doppler
Shunts evaluation - Patent Foramen Ovale | up to 72 hours
  Size will be evaluated in be viewed in subcostal view
Shunts evaluation - Patent Foramen Ovale | up to 72 hours
  Direction will be evaluated in subcostal view using color Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Rana EO Kandil, MBBCh, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt; Aly M Abdel-Mohsen, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Marwa M Farag, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt; Mohamed A Khalifa, MBBCh, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt